CLINICAL TRIAL: NCT04232553
Title: A Phase 3, Multicenter, Open-Label, Long-Term Extension Study to Evaluate the Long-Term Efficacy and Safety of Mirikizumab in Patients With Crohn's Disease
Brief Title: A Long-term Extension Study of Mirikizumab (LY3074828) in Participants With Crohn's Disease
Acronym: VIVID-2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16628; I6T-MC-AMAX (Other: Eli Lilly and Company); 2022-502841-91-00 (EU CTIS Number); 2019-002687-27 (EudraCT Number)
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Results first posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — mirikizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- AMAM Mirikizumab (Miri): Miri 300 mg SC (Experimental): Participants assigned to mirikizumab in Study AMAM who achieved Endoscopic Response at Week 52 of AMAM continued into Study AMAX and received mirikizumab 300 milligrams (mg) subcutaneously (SC) every 4 weeks (Q4W) for 52 weeks.
  Interventions: Drug: Mirikizumab
- AMAM Miri: Miri 900 mg IV Then 300 mg SC (Experimental): Participants assigned to mirikizumab in Study AMAM who did not achieve Endoscopic Response at Week 52 of AMAM continued into Study AMAX and received mirikizumab 900 mg intravenously (IV) Q4W for 3 doses, followed by mirikizumab 300 mg SC Q4W for 52 weeks.
  Interventions: Drug: Mirikizumab
- AMAM Placebo (PBO)/Miri: Miri 300 mg SC (Experimental): Participants assigned to placebo in Study AMAM who switched from placebo to mirikizumab at week 12 and achieved Endoscopic Response at Week 52 of AMAM continued into Study AMAX and received mirikizumab 300 mg SC Q4W for 52 weeks.
  Interventions: Drug: Mirikizumab
- AMAM PBO/Miri: Miri 900 mg IV Then 300 mg SC (Experimental): Participants assigned to placebo in Study AMAM who switched from placebo to mirikizumab at week 12 and did not achieve Endoscopic Response at Week 52 of AMAM continued into Study AMAX and received mirikizumab 900 mg IV Q4W for 3 doses, followed by mirikizumab 300 mg SC Q4W for 52 weeks.
  Interventions: Drug: Mirikizumab
- AMAM Ustekinumab (Uste): Miri 300 mg SC (Experimental): Participants assigned to ustekinumab in Study AMAM who achieved Endoscopic Response at Week 52 of AMAM continued into Study AMAX and received mirikizumab 300 mg SC Q4W for 52 weeks.
  Interventions: Drug: Mirikizumab
- AMAM Uste: Miri 900 mg IV Then 300 mg SC (Experimental): Participants assigned to ustekinumab in Study AMAM who did not achieve Endoscopic Response at Week 52 of AMAM continued into Study AMAX and received mirikizumab 900 mg IV Q4W for 3 doses, followed by mirikizumab 300 mg SC Q4W for 52 weeks.
  Interventions: Drug: Mirikizumab
- AMAM PBO: Miri 300 mg SC (Experimental): Participants assigned to placebo in Study AMAM who achieved Endoscopic Response at Week 52 of AMAM continued into Study AMAX and received mirikizumab 300 mg SC Q4W for 52 weeks.
  Interventions: Drug: Mirikizumab
- AMAM PBO: Miri 900 mg IV Then 300 mg SC (Experimental): Participants assigned to placebo in Study AMAM who did not achieve Endoscopic Response at Week 52 of AMAM continued into Study AMAX and received mirikizumab 900 mg IV Q4W for 3 doses, followed by mirikizumab 300 mg SC Q4W for 52 weeks.
  Interventions: Drug: Mirikizumab
- All AMAG Participants: Miri 300 mg SC (Experimental): Participants from Study AMAG who continued into Study AMAX received mirikizumab 300 mg SC Q4W for 52 weeks.
  Interventions: Drug: Mirikizumab

INTERVENTIONS:
Drug: Mirikizumab — Administered Q4W
  Other Names: LY3074828

SUMMARY:
The reason for this study is to determine the long-term efficacy and safety of the study drug mirikizumab in participants with Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have completed study I6T-MC-AMAG (NCT02891226) or study I6T-MC-AMAM (NCT03926130)
* If female, participant must meet the contraception requirements

Exclusion Criteria:

* Participants must not have developed a new condition, including cancer in the previous study (I6T-MC-AMAG or I6T-MC-AMAM) that would pose an unacceptable risk in the trial.
* Participants must not have any important infections including, but not limited to, hepatitis B, hepatitis C, HIV/AIDS, and active tuberculosis (TB) during either previous study.

Note: Participants with a history of active TB with documentation of treatment by the Centers for Disease Control (CDC) and/or World Health Organization (WHO) criteria prior to the originator study are not excluded from the study.

* Participants must not have a known hypersensitivity to any component of mirikizumab or have experienced acute systemic hypersensitivity event with previous study drug administration in the originating study that precludes mirikizumab therapy.
* Participation must not be pregnant, lactating, or planning to become pregnant while enrolled in the study or 16 weeks after receiving the last dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 996 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2024-11-28 (Actual); Study Completion 2027-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM -5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (322):
- United States (54):
  - Digestive Health Specialists, Dothan, Alabama
  - Research Solutions of Arizona, Litchfield Park, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC, Phoenix, Arizona
  - Care Access - Gilroy, Gilroy, California
  - Newport Huntington Medical Group, Huntington Beach, California
  - California Medical Research Associates, Northridge, California
  - Connecticut Clinical Research Institute, Bristol, Connecticut
  - Gastroenterology Consultants of Clearwater, Clearwater, Florida
  - Clinical Research of West Florida, Inc. (Clearwater), Clearwater, Florida
  - IHS Health Research, Kissimmee, Florida
  - Ezy Medical Research, Miami, Florida
  - Care Access - Orlando, Orlando, Florida
  - Gastroenterology Associates of Pensacola, PA, Pensacola, Florida
  - Precision Clinical Research, Sunrise, Florida
  - USF Health, Tampa, Florida
  - Alliance Clinical Research of Tampa, Tampa, Florida
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - Grand Teton Research Group, Idaho Falls, Idaho
  - Qualmedica Research, LLC, Evansville, Indiana
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - Delta Research Partners, Monroe, Louisiana
  - Capital Digestive Care - Chevy Chase, Chevy Chase, Maryland
  - Woodholme Gastroenterology Associates - Glen Burnie, Glen Burnie, Maryland
  - The Digestive Health Center of Michigan (DHCMI), Chesterfield, Michigan
  - Revive Research Institute, Inc., Farmington Hills, Michigan
  - MNGI Digestive Health - Plymouth Endoscopy Center & Clinic, Plymouth, Minnesota
  - Washington University Medical School, St Louis, Missouri
  - Care Access - Las Vegas, Las Vegas, Nevada
  - Holy Name Medical Center, Teaneck, New Jersey
  - Clinical & Translational Research Center (CTRC), Chapel Hill, North Carolina
  - Carolina Digestive Diseases and Endoscopy Center, Greenville, North Carolina
  - Care Access - Kinston, Kinston, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ohio Gastroenterology, Columbus, Ohio
  - Ohio State University, Hilliard, Ohio
  - North Shore Gastroenterology & Endoscopy Centers, Westlake, Ohio
  - The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University Gastroenterology, Providence, Rhode Island
  - Gastroenterology Associates of Orangeburg, Orangeburg, South Carolina
  - Gastroenterology Center Of The Midsouth, Cordova, Tennessee
  - First Surgical Hospital, Bellaire, Texas
  - Baylor College of Medicine Medical Center, Houston, Texas
  - West Texas Digestive Disease, Lubbock, Texas
  - Southern Star Research Institute, San Antonio, Texas
  - Tyler Research Institute, Tyler, Texas
  - Care Access - Ogden, Ogden, Utah
  - Care Access - Salt Lake City, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Clinical Research Partners, LLC, Richmond, Virginia
  - Tidewater Physicians Multispecialty Group Clinical Research, Williamsburg, Virginia
  - Washington Gastroenterology - Bellevue, Bellevue, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Washington Gastroenterology - Tacoma, Tacoma, Washington
- DOM Centro de Reumatología, Buenos Aires, Argentina
- Australia (7):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - St Vincent's Hospital, Sydney, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Coastal Digestive Health, Maroochydore, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Royal Melbourne Hospital, Parkville, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Austria (3):
  - Medizinische Universitaet Innsbruck, Innsbruck, Tyrol
  - Universitaetsklinikum Allgemeines Krankenhaus Wien, Vienna, Vienna
  - Uniklinikum Salzburg, Salzburg
- Belgium (4):
  - Imelda General Hospital, Bonheiden, Antwerpen
  - Université Libre de Bruxelles - Hôpital Erasme, Brussels, Bruxelles-Capitale, Région de
  - UZ Gent, Ghent, Oost-Vlaanderen
  - UZ Leuven, Leuven, Vlaams-Brabant
- Brazil (17):
  - CLIAGEN Clínica de Atenção em Gastroenterologia, Especialidades e Nutrição, Salvador, Estado de Bahia
  - L2IP - Instituto de Pesquisas Clínicas, Brasília, Federal District
  - Chronos Pesquisa Clínica, Brasília, Federal District
  - Hospital Felicio Rocho, Belo Horizonte, Minas Gerais
  - Fundação Universidade de Caxias do Sul (FUCS), Caxias do Sul, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Núcleo de Pesquisa Clínica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Faculdade de Medicina da UNESP, Botucatu, São Paulo
  - Centro de Pesquisa Sao Lucas, Campinas, São Paulo
  - Pesquisare Saude, Santo André, São Paulo
  - Praxis Pesquisa Medica, Santo André, São Paulo
  - Centro Multidisciplinar de Estudos Clinicos, São Bernardo do Campo, São Paulo
  - Hospital Sírio Libanês, São Paulo, São Paulo
  - CPQuali Pesquisa Clínica, São Paulo
  - Instituto de Assistência Médica ao Servidor Público Estadual - IAMSPE/HSPE-FMO Conhecer Centro de Oncolog -T, São Paulo
  - Clínica Hepatogastro JK, São Paulo
- Canada (5):
  - Gastroenterology and internal medicine research institute, Edmonton, Alberta
  - GIRI GI Research Institute - Vancouver, Vancouver, British Columbia
  - Private Practice - Dr. Bruce Musgrave, Kentville, Nova Scotia
  - Victoria Hospital, London, Ontario
  - Private Practice - Dr. Stephane M. Gauthier, North Bay, Ontario
- China (26):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Chongqing General Hospital, Chongqing, Chongqing Municipality
  - Zhongshan Hospital Affiliated to Xiamen University, Xiamen, Fujian
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Tongji Hospital Tongji Medical,Science & Technology, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Changzhou No.2 People's Hospital, Changzhou, Jiangsu
  - Jiangsu Province Hospital of Chinese Medicine, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - The Second Affiliated hospital of Zhejiang University school of medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital YuYing Childens Hospital of Wenzhou Medical university, Wenzhou, Zhejiang
  - The First Affiliated Hospital Of Fujian Medical University, Fuzhou
- Croatia (2):
  - Klinički bolnički centar Zagreb, Zagreb, City of Zagreb
  - Klinički bolnički centar Osijek, Osijek
- Czechia (15):
  - Vojenská Nemocnice Brno, Brno, Brno-město
  - Fakultni Nemocnice u sv. Anny v Brne, Brno, Brno-město
  - Hepato-Gastroenterologie HK, Hradec Králové, Hradec Králové
  - Oblastni nemocnice Nachod, Náchod, Náchod
  - MUDr. Gregar, s.r.o., Olomouc, Olomoucký kraj
  - MUDr. Radka Koskova, s.r.o., Ostrava, Ostrava Město
  - Synexus Czech, Prague, Praha 2
  - Institut Klinicke a Experimentalni Mediciny, Prague, Praha 4
  - Fakultni Thomayerova nemocnice, Prague, Praha 4
  - AXON Clinical, Prague, Praha 5
  - Fakultni nemocnice Motol, Prague, Praha 5
  - ISCARE klinické centrum, Prague, Praha 9
  - Nemocnice Tomase Bati ve Zline, Zlín, Zlín
  - PreventaMed, Olomouc
  - Masarykova Nemocnice V Usti Nad Labem, Ústí nad Labem, Ústí Nad Labem
- Gastroenterologische Praxis Balsiger, Seibold & Partner, Aalborg, North Denmark, Denmark
- France (3):
  - Chu Saint Eloi, Montpellier, Languedoc-Roussillon
  - Centre Hospitalier Régional Universitaire de Nancy - Hôpitaux de Brabois, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Centre Hospitalier Universitaire de Poitiers, Poitiers, Vienne
- Germany (12):
  - Siloah St. Trudpert Klinikum, Pforzheim, Baden-Wurttemberg
  - Universitaetsklinikum Wuerzburg, Würzburg, Bavaria
  - Synexus Clinical Research GmbH, Frankfurt am Main, Hesse
  - Siteworks GmbH - Lauterbach, Lauterbach, Hesse
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Knappschaftskrankenhaus Bottrop, Bottrop, North Rhine-Westphalia
  - Gemeinschaftspraxis Jakobeit, Wipperfürth, North Rhine-Westphalia
  - Synexus Leipzig Clinical Research Centre, Leipzig, Saxony
  - Studiengesellschaft BSF Unternehmergesellschaft, Halle, Saxony-Anhalt
  - Allgemeine Innere Medizin I, Kiel, Schleswig-Holstein
  - RED-Institut GmbH, Oldenburg in Holstein, Schleswig-Holstein
  - Tumorzentrum Nordthüringen Medizinisches Versorgungszentrum, Nordhausen, Thuringia
- Hungary (10):
  - Synexus Magyarország Kft, Gyula, Bekes County
  - Bugát Pál Kórház, Gyöngyös, Heves County
  - Szent Borbala Korhaz, Tatabánya, Komárom-Esztergom
  - Jávorszky Ödön Kórház, Vác, Pest County
  - CLINFAN Szolgáltató Kft, Szekszárd, Tolna County
  - DRC Gyógyszervizsgáló Központ, Balatonfüred, Veszprém megye
  - Békés Megyei Központi Kórház Dr. Réthy Pál Tagkórház, Békéscsaba
  - Clinexpert Kft., Budapest
  - SYNEXUS Magyarország Kft. Eü., Budapest
  - Pannónia Magánorvosi Centrum, Budapest
- India (8):
  - Gujarat Hospital - Gastro & Vascular Centre, Surat, Gujarat
  - Grant Medical Foundation - Ruby Hall Clinic, Pune, Maharashtra
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - Dayanand Medical College and Hospital, Ludhiana, Punjab
  - SR Kalla Memorial Gastro & General Hospital, Jaipur, Rajasthan
  - Apollo Speciality Hospital - Teynampet, Chennai, Tamil Nadu
  - Postgraduate Institute of Medical Education & Research, Chandigarh
- Israel (6):
  - Sheba Medical Center, Ramat Gan, Central District
  - Kaplan Medical Center, Rehovot, Central District
  - Yitzhak Shamir Medical Center, Ẕerifin, Central District
  - Shaare Zedek Medical Center, Jerusalem, Jerusalem
  - Galilee Medical Center, Nahariya, Northern District
  - Soroka Medical Center, Beersheba, Southern District
- Italy (3):
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - IRCCS Policlinico San Donato, Milan, Milano
  - Ospedale Di Circolo, Rho, Milano
- Japan (26):
  - National Hospital Organization Hirosaki General Medical Center, Hirosaki, Aomori
  - Tsujinaka Hospital - Kashiwanoha, Kashiwa, Chiba
  - Kitakyushu Municipal Medical Center, Kitakyusyu-shi, Fukoka
  - Fukuoka University Chikushi Hospital, Chikushino-shi, Fukuoka
  - Kiryu Kosei General Hospital, Kiryū, Gunma
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital, Chuo-ku, Sapporo-shi, Hokkaido
  - Tokushukai Sapporo Tokushukai Hospital, Sapporo, Hokkaido
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Sapporo Higashi Tokushukai Hospital, Sapporo, Hokkaido
  - Hyogo College of Medicine, Nishinomiya, Hyōgo
  - Ibaraki Prefectural Central Hospital, Kasama, Ibaraki
  - Ofuna Central Hospital, Kamakura, Kanagawa
  - Mie University Hospital, Tsu, Mie-ken
  - Takagi Clinic - Sendai, Sendai, Miyagi
  - Matsuda Hospital, Hamamatsu, Shizuoka
  - Institute of Science Tokyo Hospital, Bunkyo, Tokyo
  - Kyorin University Hospital, Mitaka, Tokyo
  - Center Hospital of the National Center for Global Health and Medicine, Shinjyuku-ku, Tokyo
  - Fukuoka University Hospital, Fukuoka
  - Kagoshima University Hospital, Kagoshima
  - Sameshima Hospital, Kagoshima
  - Kumamoto University Hospital, Kumamoto
  - University Hospital,Kyoto Prefectural University of Medicine, Kyoto
  - Okayama Saiseikai Outpatient Center Hospital, Okayama
  - Tokyo Yamate Medical Center, Tokyo
  - Toyama Prefectural Central Hospital, Toyama
- Pauls Stradins Clinical Univeristy Hospital, Riga, Rīga, Latvia
- Hospital of Lithuanian University of Health Sciences Kaunas, Kaunas, Lithuania
- Mexico (4):
  - Christus Muguerza Hospital Sur, Monterrey, Nuevo León
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - Centro de Alta Especialidad en Reumatologia e Investigación del Potosi,S.C, San Luis Potosí City, San Luis Potosí
  - Scientia Investigacion Clinica S.C., Chihuahua City
- Netherlands (2):
  - Elisabeth-TweeSteden Ziekenhuis, Tilburg, North Brabant
  - Amsterdam UMC, locatie VUmc, Amsterdam, North Holland
- Poland (24):
  - Synexus Polska Sp. z o.o. Oddzial w Poznaniu, Poznan, Greater Poland Voivodeship
  - Centrum Medyczne "Medis" Manermed, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Topolowa Medicenter, Krakow, Lesser Poland Voivodeship
  - NZOZ Formed, Wadowice, Lesser Poland Voivodeship
  - Dc-Med, Swidnica, Lower Silesian Voivodeship
  - Melita Medical, Wroclaw, Lower Silesian Voivodeship
  - Reumatop, Wroclaw, Lower Silesian Voivodeship
  - Synexus - Wroclaw, Wroclaw, Lower Silesian Voivodeship
  - ZOZ Gastromed, Lublin, Lublin Voivodeship
  - ETG Zamość, Zamość, Lublin Voivodeship
  - Centrum Zdrowia MDM, Warsaw, Masovian Voivodeship
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw, Masovian Voivodeship
  - Private Practice - Dr. Korczowski Bartosz, Rzeszów, Podkarpackie Voivodeship
  - Centrum Medyczne MEDYK, Rzeszów, Podkarpackie Voivodeship
  - Nova Reuma Domyslawska i Rusilowicz Spolka Partnerska Lekarza Reumatologa i Fizjoterapeuty, Bialystok, Podlaskie Voivodeship
  - Synexus Polska Gdansku, Gdansk, Pomeranian Voivodeship
  - Synexus Polska Sp. z o.o. Oddzial w Gdyni, Gdynia, Pomeranian Voivodeship
  - Endoskopia Sp. z.o.o., Sopot, Pomeranian Voivodeship
  - Synexus Polska Sp. z o.o. Oddzial w Czestochowie, Częstochowa, Silesian Voivodeship
  - Synexus Polska - Katowicach, Katowice, Silesian Voivodeship
  - Kiepury Clinic, Sosnowiec, Silesian Voivodeship
  - NZOZ TwojeZdrowie, Elblag, Warmian-Masurian Voivodeship
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin, West Pomeranian Voivodeship
  - SONOMED Centrum Medyczne, Szczecin, West Pomeranian Voivodeship
- Romania (6):
  - Spitalul de Oncologie Monza, Bucharest, București
  - Delta Health Care, Bucharest, București
  - S.C. Centrul Medical Medicum SRL, Bucharest, București
  - Spitalul Clinic Colentina, Bucharest, București
  - S.C Centrul de Gastroenterologie Dr. Goldis S.R.L, Timișoara, Timiș County
  - Gastromed S.R.L., Constanța
- Russia (18):
  - Poliklinika Agmu "Konsul'tativno-Diagnosticheskiy Tsentr", Barnaul, Altayskiy Kray
  - Scientific Centre of Reconstructive and Restorative Surgery, Irkutsk, Irkutsk Oblast
  - Karelia Republican Hospital V.A. Baranova, Petrozavodsk, Kareliya, Respublika
  - SIH Kemerovo Regional Clinical Hosptial, Kemerovo, Kemerovo Oblast
  - Olla-Med, Moscow, Moscow
  - Nizhny Novgorod Regional Hospital N.A. Semashko, Nizhny Novgorod, Nizhny Novgorod Oblast
  - LLC "Medicine Center SibNovoMed", Novosibirsk, Novosibirsk Oblast
  - Research Institute of Physiology and Fundamental Medicine, Novosibirsk, Novosibirsk Oblast
  - Clinic of Omsk State Medical University, Omsk, Omsk Oblast
  - Rostov State Medical University, Rostov-on-Don, Rostov Oblast
  - NonState Healthcare Institution Central Clinical Hospital, Samara, Samara Oblast
  - LLC Medical Center Reavita Med SPb, Saint Petersburg, Sankt-Peterburg
  - Balt Med Clinic, Saint Petersburg, Sankt-Peterburg
  - Saint-Petersburg City Hospital of Saint Elizabeth, Saint Petersburg, Sankt-Peterburg
  - Scientific research center ECO-security, Saint Petersburg, Sankt-Peterburg
  - First Pavlov State Medical University of Saint Petersburg, Saint Petersburg, Sankt-Peterburg
  - Saint Petersburg State Budgetary Healthcare Institution City Clinical Hospital No.31, Saint Petersburg, Sankt-Peterburg
  - LLC MA New Hospital, Yekaterinburg, Sverdlovsk Oblast
- Serbia (3):
  - Clinical Hospital Center Zvezdara, Belgrade, Beograd
  - University Medical Center "Bezanijska kosa", Belgrade, Beograd
  - General Hospital "Djordje Joanovic", Zrenjanin, Vojvodina
- Slovakia (5):
  - Fakultna nemocnica s poliklinikou F.D.Roosevelta Banska Bystrica, Banská Bystrica, Banská Bystrica Region
  - Cliniq s.r.o., Bratislava, Bratislava Region
  - Gastromedic, Nové Zámky, Nitra Region
  - Gastro LM, Prešov, Presov
  - Endomed, s.r.o., Vranov N. Toplou, Presov
- South Korea (16):
  - Yonsei University-Wonju Severance Christian Hospital, Wŏnju, Kang-won-do
  - Korea University Ansan Hospital, Ansan-si, Kyǒnggi-do
  - Hanyang University Guri Hospital, Guri-si, Kyǒnggi-do
  - Ajou University Hospital, Suwon, Kyǒnggi-do
  - Yeungnam Univeristy Medical Center, Gyeongsan-si, Kyǒngsangbuk-do
  - Dong-A University Hospital, Busan, Pusan-Kwangyǒkshi
  - Inje University Haeundae Paik Hospital, Haeundae-gu, Pusan-Kwangyǒkshi
  - Chungang University Hospital, Dongjak-gu, Seoul-teukbyeolsi [Seoul]
  - Kyung Hee University Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Kangbuk Samsung Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Keimyung University Dongsan Hospital, Daegu, Taegu-Kwangyǒkshi
  - Kyungpook National University Chilgok Hospital, Deagu, Taegu-Kwangyǒkshi
  - Kyungpook National University Hospital, Junggu, Taegu-Kwangyǒkshi
  - The Catholic University of Korea, Daejeon St. Mary's Hospital, Daejeon, Taejǒn-Kwangyǒkshi
- Switzerland (3):
  - Gastroenterologische Praxis Balsiger, Seibold & Partner, Bern, Canton of Bern
  - Cantonal Hospital St.Gallen, Sankt Gallen, Canton of St. Gallen
  - Inselspital Bern, Bern
- Turkey (Türkiye) (14):
  - Eskisehir Osmangazi University, Eskişehir, Eskişehir
  - Istanbul Universitesi Cerrahpasa, Istanbul- Fatih, Istanbul
  - Dokuz Eylül Üniversitesi, Balçova, İzmir
  - Kocaeli University Medical Faculty Hospital, İzmit, Kocaeli
  - Ankara City Hospital, Ankara
  - Hacettepe Universite Hastaneleri, Ankara
  - Gazi University Health Research and Application Center Gazi Hospital, Ankara
  - Antalya Egitim ve Arastırma Hastanesi, Antalya
  - Uludag Universitesi, Bursa
  - Trakya University, Edirne
  - Mustafa Kemal Universitesi, Hatay
  - Medicana Kadiköy Hastanesi, Istanbul
  - Acbadem Kozyatagi Hospital, Istanbul
  - Mersin University, Mersin
- Ukraine (19):
  - Medical Center Family Medicine Clinic, Dnipro, Dnipropetrovsk Oblast
  - Communal non-profit enterprise "Regional clinical hospital of Ivano-Frankivsk Regional Council", Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - City Clinical Hospital No. 2, Kharkiv, Kharkivs’ka Oblast’
  - Medbud Clinic, Kyiv, Kyivska Oblast
  - University Hospital branch of Danylo Halytsky Lviv National Medical University (UH DHLNMU), Lviv, Lviv Oblast
  - Municipal non-profit enterprise'Odesa Regional Clinical Hospital'of Odesa Regional Council, Odesa, Odesa Oblast
  - City Clinical Hospital #1, Vinnitsya National Medical University, Vinnytsia, Vinnytsia Oblast
  - Medical Clinical Investigational Center of Medical Center Health Clinic, Vinnytsia, Vinnytsia Oblast
  - Municipal Nonprofit Enterprise "Vinnytsia Regional Clinical Hospital n.a. M. I. Pyrohov of Vinnytsia Regio -T, Vinnytsia, Vinnytsia Oblast
  - VNMU, Vinnytsia, Vinnytsia Oblast
  - Transcarpathian Regional Hospital im.Andriya Novak, Uzhhorod, Zakarpattia Oblast
  - Communal Non-profit Enterprise "City Hospital #6" of Zaporizhzhia City Council, Zaporizhia, Zaporizhzhia Oblast
  - Diacenter, Zaporizhzhia, Zaporizhzhia Oblast
  - Chernivtsi Regional Clinical Hospital, Chernivtsi
  - Medical Center Ok!Clinic+, Kyiv
  - Kyiv Railway Clinical Hospital No.2 of Branch Health Center of the Public Joint Stock Company Ukrainian Ra -T, Kyiv
  - Medical Center of Limited Liability Company "Medical Center "Consilium Medical", Kyiv
  - Municipal non-profit enterprise of Kyiv Regional Council "Kyiv Regional Center for Rehabilitation Medicine", Kyiv
  - Municipal Nonprofit Enterprise of Kyiv Region Council "Kyiv Regional Clinical Hospital", Kyiv
- United Kingdom (3):
  - Addenbrooke's Hospital, Cambridge, Cambridgeshire
  - Whipps Cross University Hospital, London, England
  - Synexus Wales Clinical Research Centre, Cardiff

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Long-term Extension Study of Mirikizumab (LY3074828) in Participants With Crohn's Disease — https://trials.lilly.com/en-US/trial/244316

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligibility for Study I6T-MC-AMAX (AMAX; NCT04232553) required completion of one of the originating studies: either Study I6T-MC-AMAM (AMAM; NCT03926130) or Study I6T-MC-AMAG (AMAG; NCT02891226). Participants from Study AMAM were classified as having achieved Endoscopic Response if they achieved a reduction from baseline in the Simple Endoscopic Score for Crohn's Disease [SES-CD] total score of greater than or equal to (>=) 50% at Week 52.
Pre-assignment Details: (continued) Participants from Study AMAM were classified as not having achieved Endoscopic Response if they did not achieve a reduction from baseline in SES-CD total score >= 50% at Week 52.
Period: Overall Study
Arm/Group | AMAM Mirikizumab (Miri): Miri 300 mg SC | AMAM Miri: Miri 900 mg IV Then 300 mg SC | AMAM Placebo (PBO)/Miri: Miri 300 mg SC | AMAM PBO/Miri: Miri 900 mg IV Then 300 mg SC | AMAM Ustekinumab (Uste): Miri 300 mg SC | AMAM Uste: Miri 900 mg IV Then 300 mg SC | AMAM PBO: Miri 300 mg SC | AMAM PBO: Miri 900 mg IV Then 300 mg SC | All AMAG Participants: Miri 300 mg SC
Started | 287 | 222 | 29 | 34 | 138 | 109 | 18 | 53 | 106
Received at Least One Dose of Study Drug | 287 | 222 | 29 | 34 | 138 | 109 | 18 | 53 | 106
Completed (Participants who completed the 52-week treatment were considered as 'completed'.) | 275 | 209 | 28 | 31 | 133 | 106 | 18 | 51 | 104
Not Completed | 12 | 13 | 1 | 3 | 5 | 3 | 0 | 2 | 2
Not completed — Adverse Event | 3 | 2 | 1 | 2 | 1 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Other - As reported by the investigator | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 5 | 0 | 0 | 2 | 2 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- AMAM Miri: Miri 300 mg SC: Participants assigned to mirikizumab in Study AMAM who achieved Endoscopic Response at Week 52 of AMAM continued into Study AMAX and received mirikizumab 300 mg SC Q4W for 52 weeks.
- AMAM Miri: Miri 900 mg IV Then 300 mg SC: Participants assigned to mirikizumab in Study AMAM who did not achieve Endoscopic Response at Week 52 of AMAM continued into Study AMAX and received mirikizumab 900 mg IV Q4W for 3 doses, followed by mirikizumab 300 mg SC Q4W for 52 weeks.
- AMAM PBO/Miri: Miri 300 mg SC: Participants assigned to placebo in Study AMAM who switched from placebo to mirikizumab at week 12 and achieved Endoscopic Response at Week 52 of AMAM continued into Study AMAX and received mirikizumab 300 mg SC Q4W for 52 weeks.
- AMAM Uste: Miri 300 mg SC: Participants assigned to ustekinumab in Study AMAM who achieved Endoscopic Response at Week 52 of AMAM continued into Study AMAX and received mirikizumab 300 mg SC Q4W for 52 weeks.
- Total: Total of all reporting groups
Arm/Group | AMAM Miri: Miri 300 mg SC | AMAM Miri: Miri 900 mg IV Then 300 mg SC | AMAM PBO/Miri: Miri 300 mg SC | AMAM PBO/Miri: Miri 900 mg IV Then 300 mg SC | AMAM Uste: Miri 300 mg SC | AMAM Uste: Miri 900 mg IV Then 300 mg SC | AMAM PBO: Miri 300 mg SC | AMAM PBO: Miri 900 mg IV Then 300 mg SC | All AMAG Participants: Miri 300 mg SC | Total
Number analyzed (Participants) | 287 | 222 | 29 | 34 | 138 | 109 | 18 | 53 | 106 | 996
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (12.84) | 38.4 (13.66) | 39.5 (16.00) | 37.7 (11.92) | 39.2 (12.84) | 37.6 (12.68) | 37.6 (9.52) | 38.0 (12.88) | 41.5 (12.20) | 38.4 (12.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 88 | 17 | 11 | 70 | 54 | 7 | 21 | 49 | 441
  Male | 163 | 134 | 12 | 23 | 68 | 55 | 11 | 32 | 57 | 555
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 6
  Asian | 68 | 61 | 7 | 5 | 31 | 21 | 3 | 6 | 13 | 215
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 5 | 0 | 1 | 3 | 3 | 0 | 0 | 7 | 23
  White | 207 | 154 | 21 | 26 | 102 | 84 | 14 | 45 | 85 | 738
  More than one race | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 4
  Unknown or Not Reported | 5 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Australia | 3 | 4 | 0 | 1 | 0 | 0 | 0 | 4 | 1 | 13
  Austria | 1 | 5 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 9
  Belgium | 2 | 3 | 0 | 1 | 0 | 1 | 0 | 1 | 3 | 11
  Brazil | 14 | 11 | 0 | 3 | 7 | 7 | 2 | 3 | 0 | 47
  Canada | 11 | 4 | 4 | 0 | 5 | 3 | 1 | 1 | 0 | 29
  China | 34 | 32 | 5 | 4 | 10 | 16 | 0 | 4 | 0 | 105
  Croatia | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
  Czechia | 12 | 14 | 5 | 2 | 8 | 7 | 2 | 2 | 6 | 58
  France | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
  Germany | 15 | 4 | 1 | 0 | 2 | 5 | 2 | 2 | 0 | 31
  Hungary | 10 | 3 | 1 | 1 | 5 | 5 | 1 | 1 | 4 | 31
  India | 4 | 6 | 1 | 0 | 5 | 1 | 0 | 0 | 0 | 17
  Israel | 3 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 8
  Italy | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
  Japan | 6 | 5 | 0 | 1 | 9 | 2 | 0 | 1 | 13 | 37
  Latvia | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
  Lithuania | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 4
  Mexico | 3 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 7
  Netherlands | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 5 | 8
  Poland | 40 | 33 | 0 | 4 | 17 | 22 | 2 | 8 | 16 | 142
  Romania | 5 | 5 | 0 | 0 | 1 | 1 | 1 | 0 | 4 | 17
  Russia | 18 | 18 | 2 | 5 | 11 | 5 | 1 | 8 | 6 | 74
  Serbia | 4 | 1 | 4 | 2 | 3 | 2 | 0 | 2 | 0 | 18
  Slovakia | 3 | 4 | 0 | 0 | 3 | 3 | 0 | 1 | 0 | 14
  South Korea | 21 | 17 | 1 | 0 | 6 | 2 | 3 | 1 | 0 | 51
  Switzerland | 2 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 6
  Turkey | 15 | 9 | 1 | 1 | 1 | 5 | 0 | 2 | 0 | 34
  Ukraine | 22 | 11 | 2 | 3 | 18 | 11 | 2 | 1 | 13 | 83
  United Kingdom | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  United States | 26 | 26 | 1 | 3 | 19 | 7 | 1 | 6 | 35 | 124

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Endoscopic Response at Week 52 (Participants Originating From AMAM Study)
Description: Endoscopic Response defined as ≥50% reduction from AMAM study baseline in Simple Endoscopic Score for Crohn's Disease (SES-CD) total score. The SES-CD evaluates 4 endoscopic variables (presence/size of ulcers, extent of ulcerated surface, extent of affected surface, and presence/severity of stenosis) across 5 ileocolonic bowel segments (ileum, right colon, transverse colon, left colon, and rectum), with each of the 4 variables scored from 0 (best) to 3 (worst) per segment, resulting in 20 individual assessments. Total SES-CD score is the sum of all 20 individual assessment scores across all the bowel segments. Scores range from 0 to 56, with higher scores indicating more severe disease.
Time Frame: Week 52
Population: All enrolled participants originating from the AMAM study who received at least one dose of study drug and had a baseline SES-CD total score ≥7 (or ≥4 for isolated ileal disease) in the AMAM study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AMAM Miri: Miri 300 mg SC | AMAM Miri: Miri 900 mg IV Then 300 mg SC | AMAM PBO/Miri: Miri 300 mg SC | AMAM PBO/Miri: Miri 900 mg IV Then 300 mg SC | AMAM Uste: Miri 300 mg SC | AMAM Uste: Miri 900 mg IV Then 300 mg SC | AMAM PBO: Miri 300 mg SC | AMAM PBO: Miri 900 mg IV Then 300 mg SC
Number analyzed (Participants) | 269 | 195 | 28 | 31 | 132 | 97 | 18 | 49
percentage of participants | 82.1 [77.4 to 86.8] | 29.7 [23.0 to 36.4] | 92.6 [82.7 to 100] | 38.7 [23.7 to 56.2] | 75.0 [67.3 to 82.7] | 39.7 [29.6 to 49.8] | 94.1 [82.6 to 100] | 51.4 [36.9 to 65.8]

2. Primary Outcome: Percentage of Participants Achieving Clinical Remission at Week 52 (Participants Originating From AMAM Study)
Description: Clinical remission was defined as a Crohn's Disease Activity Index (CDAI) total score < (less than) 150. The CDAI measures the severity of active disease using 8 disease variables: stool frequency, severity of abdominal pain, degree of general well-being, presence or absence of extra-intestinal manifestations, presence or absence of fistula, use or non-use of antidiarrheal agents, presence or absence of an abdominal mass, hematocrit, and body weight. Each variable is assigned a specific weight/multiplier, and the weighted values are summed to produce a CDAI total score. CDAI total scores can range from 0 to 600, with higher scores indicating more severe disease.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AMAM Miri: Miri 300 mg SC | AMAM Miri: Miri 900 mg IV Then 300 mg SC | AMAM PBO/Miri: Miri 300 mg SC | AMAM PBO/Miri: Miri 900 mg IV Then 300 mg SC | AMAM Uste: Miri 300 mg SC | AMAM Uste: Miri 900 mg IV Then 300 mg SC | AMAM PBO: Miri 300 mg SC | AMAM PBO: Miri 900 mg IV Then 300 mg SC
Number analyzed (Participants) | 269 | 195 | 28 | 31 | 132 | 97 | 18 | 49
percentage of participants | 79.2 [74.1 to 84.4] | 65.9 [58.8 to 72.9] | 76.6 [60.1 to 93.2] | 55.9 [37.6 to 74.2] | 75.8 [67.9 to 83.6] | 74.6 [65.2 to 84.0] | 84.9 [65.3 to 100] | 68.5 [53.8 to 83.1]

3. Secondary Outcome: Percentage of Participants Achieving Alternate Endoscopic Remission at Week 52 (Participants Originating From AMAM Study)
Description: Alternate endoscopic remission is defined as SES-CD Total Score ≤4 with at least a 2-point reduction from the AMAM study baseline and no subscore >1. The SES-CD evaluates 4 endoscopic variables (presence/size of ulcers, extent of ulcerated surface, extent of affected surface, and presence/severity of stenosis) across 5 ileocolonic bowel segments (ileum, right colon, transverse colon, left colon, and rectum), with each of the 4 variables scored from 0 (best) to 3 (worst) per segment, resulting in 20 individual assessments. Total SES-CD score is the sum of all 20 individual assessment scores across all the bowel segments. Scores range from 0 to 56, with higher scores indicating more severe disease. No subscore >1 is defined as no individual assessment score >1 across all 20 individual assessments.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AMAM Miri: Miri 300 mg SC | AMAM Miri: Miri 900 mg IV Then 300 mg SC | AMAM PBO/Miri: Miri 300 mg SC | AMAM PBO/Miri: Miri 900 mg IV Then 300 mg SC | AMAM Uste: Miri 300 mg SC | AMAM Uste: Miri 900 mg IV Then 300 mg SC | AMAM PBO: Miri 300 mg SC | AMAM PBO: Miri 900 mg IV Then 300 mg SC
Number analyzed (Participants) | 269 | 195 | 28 | 31 | 132 | 97 | 18 | 49
percentage of participants | 54.6 [48.4 to 60.7] | 14.2 [9.1 to 19.3] | 66.3 [48.0 to 84.5] | 25.8 [13.7 to 43.2] | 47.1 [38.3 to 56.0] | 22.1 [13.5 to 30.6] | 63.1 [39.6 to 86.6] | 32.6 [19.0 to 46.1]

4. Secondary Outcome: Percentage of Participants Achieving Clinical Response by Patient Reported Outcome (PRO) at Week 52 - (Participants Originating From AMAM Study)
Description: Clinical response by Patient Reported Outcome (PRO) was defined as a ≥30% decrease from baseline in stool frequency (SF) and/or abdominal pain (AP) score, with neither symptom worsening from baseline. SF was measured as the number of liquid or very soft stools per day. AP was scored daily on a 4-point scale: 0 = none, 1 = mild, 2 = moderate, and 3 = severe.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AMAM Miri: Miri 300 mg SC | AMAM Miri: Miri 900 mg IV Then 300 mg SC | AMAM PBO/Miri: Miri 300 mg SC | AMAM PBO/Miri: Miri 900 mg IV Then 300 mg SC | AMAM Uste: Miri 300 mg SC | AMAM Uste: Miri 900 mg IV Then 300 mg SC | AMAM PBO: Miri 300 mg SC | AMAM PBO: Miri 900 mg IV Then 300 mg SC
Number analyzed (Participants) | 269 | 195 | 28 | 31 | 132 | 97 | 18 | 49
percentage of participants | 87.3 [83.1 to 91.4] | 74.7 [68.4 to 81.0] | 88.9 [76.8 to 100] | 63.3 [45.7 to 81.0] | 86.2 [80.1 to 92.3] | 84.0 [76.6 to 91.5] | 97.8 [86.4 to 100] | 78.2 [66.0 to 90.3]

5. Secondary Outcome: Fecal Calprotectin at Week 12 (Participants Originating From AMAM Study)
Description: Fecal calprotectin is an indicator of inflammation in the intestines with higher levels indicative of higher levels of inflammation.
Time Frame: Week 12
Population: All enrolled participants originating from the AMAM study who received at least one dose of study drug and had a baseline SES-CD total score ≥7 (or ≥4 for isolated ileal disease) in the AMAM study, and had evaluable fecal calprotectin data.
Measure: Median (Inter-Quartile Range); unit: micrograms per gram (μg/g)
Arm/Group | AMAM Miri: Miri 300 mg SC | AMAM Miri: Miri 900 mg IV Then 300 mg SC | AMAM PBO/Miri: Miri 300 mg SC | AMAM PBO/Miri: Miri 900 mg IV Then 300 mg SC | AMAM Uste: Miri 300 mg SC | AMAM Uste: Miri 900 mg IV Then 300 mg SC | AMAM PBO: Miri 300 mg SC | AMAM PBO: Miri 900 mg IV Then 300 mg SC
Number analyzed (Participants) | 230 | 169 | 27 | 27 | 111 | 82 | 13 | 42
micrograms per gram (μg/g) | 110.5 [37.0 to 293.0] | 310.0 [104.0 to 962.0] | 134.0 [15.0 to 484.0] | 168.0 [62.0 to 761.0] | 113.0 [40.0 to 364.0] | 312.5 [85.0 to 834.0] | 46.0 [15.0 to 415.0] | 333.5 [67.0 to 984.0]

6. Secondary Outcome: C-Reactive Protein (CRP) at Week 12 (Participants Originating From AMAM Study)
Description: C-Reactive Protein is a biomarker of systemic inflammation measured in the blood, with elevated levels indicating increased inflammatory activity in the body.
Time Frame: Week 12
Population: All enrolled participants originating from the AMAM study who received at least one dose of study drug and had a baseline SES-CD total score ≥7 (or ≥4 for isolated ileal disease) in the AMAM study, and had evaluable C-Reactive Protein data.
Measure: Median (Inter-Quartile Range); unit: milligram per liter (mg/L)
Arm/Group | AMAM Miri: Miri 300 mg SC | AMAM Miri: Miri 900 mg IV Then 300 mg SC | AMAM PBO/Miri: Miri 300 mg SC | AMAM PBO/Miri: Miri 900 mg IV Then 300 mg SC | AMAM Uste: Miri 300 mg SC | AMAM Uste: Miri 900 mg IV Then 300 mg SC | AMAM PBO: Miri 300 mg SC | AMAM PBO: Miri 900 mg IV Then 300 mg SC
Number analyzed (Participants) | 264 | 183 | 28 | 28 | 127 | 93 | 15 | 46
milligram per liter (mg/L) | 1.4 [0.6 to 4.6] | 2.7 [1.1 to 5.4] | 1.4 [1.0 to 5.0] | 3.2 [1.1 to 6.2] | 1.3 [0.6 to 3.8] | 3.5 [0.9 to 6.8] | 2.3 [0.4 to 4.7] | 3.7 [1.3 to 7.3]

7. Secondary Outcome: Change From Baseline in Health Related Quality of Life at Week 52 : Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score (Participants Originating From AMAM Study)
Description: The Inflammatory Bowel Disease Questionnaire (IBDQ) is a 32-item participant completed questionnaire that measures 4 aspects of patients' lives: symptoms directly related to the primary bowel disturbance (10 items), systemic symptoms (5 items), emotional function (12 items), and social function(5 items). Responses are graded on a 7-point Likert scale in which 7 denotes "not a problem at all" and 1 denotes "a very severe problem." IBDQ total score is calculated as the sum of all questions. Total scores range from 32 to 224; a higher score indicates a better quality of life.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AMAM Miri: Miri 300 mg SC | AMAM Miri: Miri 900 mg IV Then 300 mg SC | AMAM PBO/Miri: Miri 300 mg SC | AMAM PBO/Miri: Miri 900 mg IV Then 300 mg SC | AMAM Uste: Miri 300 mg SC | AMAM Uste: Miri 900 mg IV Then 300 mg SC | AMAM PBO: Miri 300 mg SC | AMAM PBO: Miri 900 mg IV Then 300 mg SC
Number analyzed (Participants) | 269 | 195 | 28 | 31 | 132 | 97 | 18 | 49
score on a scale | 57.3 (1.99) | 46.1 (2.32) | 47.4 (6.12) | 38.6 (5.81) | 50.5 (2.82) | 49.9 (3.29) | 65.3 (7.84) | 46.4 (4.62)

ADVERSE EVENTS:
Time Frame: Baseline Up to Week 52
Description: * All enrolled participants who received at least one dose of study drug. As pre-specified in the statistical analysis plan (SAP), adverse events were reported by treatment regimen.
  * Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | AMAM Miri: Miri 300 mg SC | AMAM Miri: Miri 900 mg IV Then 300 mg SC | AMAM PBO/Miri: Miri 300 mg SC | AMAM PBO/Miri: Miri 900 mg IV Then 300 mg SC | AMAM Uste: Miri 300 mg SC | AMAM Uste: Miri 900 mg IV Then 300 mg SC | AMAM PBO: Miri 300 mg SC | AMAM PBO: Miri 900 mg IV Then 300 mg SC | All AMAG Participants: Miri 300 mg SC
All-Cause Mortality (participants affected / at risk) | 0/287 | 1/222 | 0/29 | 1/34 | 0/138 | 0/109 | 0/18 | 0/53 | 0/106
Serious Adverse Events (participants affected / at risk) | 19/287 | 20/222 | 1/29 | 8/34 | 9/138 | 9/109 | 0/18 | 7/53 | 3/106
Other Adverse Events (participants affected / at risk) | 189/287 | 138/222 | 16/29 | 21/34 | 82/138 | 69/109 | 12/18 | 33/53 | 68/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | AMAM Miri: Miri 300 mg SC (N=287) | AMAM Miri: Miri 900 mg IV Then 300 mg SC (N=222) | AMAM PBO/Miri: Miri 300 mg SC (N=29) | AMAM PBO/Miri: Miri 900 mg IV Then 300 mg SC (N=34) | AMAM Uste: Miri 300 mg SC (N=138) | AMAM Uste: Miri 900 mg IV Then 300 mg SC (N=109) | AMAM PBO: Miri 300 mg SC (N=18) | AMAM PBO: Miri 900 mg IV Then 300 mg SC (N=53) | All AMAG Participants: Miri 300 mg SC (N=106)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Ileal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Terminal ileitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial translocation (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial paresis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intrusive thoughts (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Schizoaffective disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0/124 (0) | 0/88 (0) | 0/17 (0) | 0/11 (0) | 1/70 (1) | 0/54 (0) | 0/7 (0) | 0/21 (0) | 0/49 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 1/124 (1) | 0/88 (0) | 0/17 (0) | 0/11 (0) | 0/70 (0) | 0/54 (0) | 0/7 (0) | 0/21 (0) | 0/49 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | AMAM Miri: Miri 300 mg SC (N=287) | AMAM Miri: Miri 900 mg IV Then 300 mg SC (N=222) | AMAM PBO/Miri: Miri 300 mg SC (N=29) | AMAM PBO/Miri: Miri 900 mg IV Then 300 mg SC (N=34) | AMAM Uste: Miri 300 mg SC (N=138) | AMAM Uste: Miri 900 mg IV Then 300 mg SC (N=109) | AMAM PBO: Miri 300 mg SC (N=18) | AMAM PBO: Miri 900 mg IV Then 300 mg SC (N=53) | All AMAG Participants: Miri 300 mg SC (N=106)
Anaemia (Blood and lymphatic system disorders) | 10 (10) | 4 (6) | 1 (1) | 3 (3) | 7 (8) | 4 (4) | 1 (2) | 2 (2) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (4) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 3 (3) | 5 (7) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Birth mark (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gilbert's syndrome (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0/163 (0) | 0/134 (0) | 0/12 (0) | 0/23 (0) | 1/68 (1) | 0/55 (0) | 0/11 (0) | 0/32 (0) | 0/57 (0)
Type v hyperlipidaemia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Androgen deficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polycystic ovarian syndrome (Endocrine disorders) | 0/124 (0) | 1/88 (1) | 0/17 (0) | 0/11 (0) | 0/70 (0) | 0/54 (0) | 0/7 (0) | 0/21 (0) | 0/49 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chorioretinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dacryoadenitis acquired (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macular degeneration (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Panophthalmitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital swelling (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scleritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 8 (8) | 9 (11) | 1 (1) | 1 (2) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 4 (5)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 11 (13) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorectal polyp (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (5) | 5 (6) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Crohn's disease (Gastrointestinal disorders) | 2 (2) | 4 (4) | 2 (2) | 1 (1) | 3 (3) | 7 (7) | 1 (2) | 2 (2) | 2 (2)
Dental caries (Gastrointestinal disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 9 (9) | 0 (0) | 0 (0) | 2 (2) | 4 (5) | 2 (2) | 0 (0) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (4)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Erosive oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival recession (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 5 (5) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperchlorhydria (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inflammatory bowel disease (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Large intestine erosion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (4) | 4 (4) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Reflux gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Terminal ileitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 6 (7) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Adverse drug reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Application site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Application site pain (General disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cyst (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug intolerance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye complication associated with device (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (4) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 4 (4) | 3 (3)
Influenza like illness (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion site oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site dermatitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site discharge (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 2 (7) | 1 (1) | 0 (0) | 0 (0) | 2 (15) | 0 (0) | 0 (0) | 0 (0) | 3 (28)
Injection site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site hypersensitivity (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site inflammation (General disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 5 (46) | 1 (19) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (27)
Injection site pruritus (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 2 (6) | 2 (3) | 0 (0) | 0 (0) | 5 (31) | 3 (4) | 0 (0) | 0 (0) | 2 (8)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Mass (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pseudopolyp (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 6 (9) | 9 (10) | 1 (1) | 2 (2) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 5 (6)
Secretion discharge (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tenderness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Xerosis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis sclerosing (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Allergy to animal (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 2 (3) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related hypersensitivity reaction (Immune system disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Type ii hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Cellulitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronavirus pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 35 (39) | 25 (26) | 2 (2) | 2 (2) | 12 (12) | 14 (14) | 5 (5) | 7 (7) | 12 (12)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema infected (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 6 (9) | 4 (5) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 2 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Hiv infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected bite (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 6 (7) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Labyrinthitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Latent tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 19 (22) | 0 (0) | 2 (2) | 0 (0) | 7 (7) | 5 (6) | 2 (3) | 5 (7) | 6 (7)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericoronitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulpitis dental (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotavirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salpingo-oophoritis (Infections and infestations) | 0/124 (0) | 0/88 (0) | 0/17 (0) | 0/11 (0) | 0/70 (0) | 1/54 (2) | 0/7 (0) | 0/21 (0) | 0/49 (0)
Scabies (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sexually transmitted disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 6 (7) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 2 (2) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suspected covid-19 (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea cruris (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea manuum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 14 (18) | 16 (20) | 2 (3) | 1 (1) | 7 (7) | 5 (5) | 1 (2) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 4 (5) | 4 (4) | 1 (1) | 1 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 4 (5) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Viral pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0/124 (0) | 1/88 (1) | 0/17 (0) | 1/11 (1) | 0/70 (0) | 0/54 (0) | 0/7 (0) | 0/21 (0) | 0/49 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0/124 (0) | 0/88 (0) | 0/17 (0) | 0/11 (0) | 0/70 (0) | 0/54 (0) | 0/7 (0) | 0/21 (0) | 1/49 (1)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Animal scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chemical burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foreign body in throat (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Immunisation reaction (Injury, poisoning and procedural complications) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mallet finger (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural site reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scapula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (3) | 4 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alpha tumour necrosis factor increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Antinuclear antibody positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ast/alt ratio abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biopsy breast (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood bicarbonate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood calcium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood cholesterol decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 3 (3) | 2 (3) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 8 (10) | 6 (6) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood folate decreased (Investigations) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood iron decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Blood triglycerides increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatitis b dna assay positive (Investigations) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
High density lipoprotein decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interleukin level increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Low density lipoprotein increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 4 (6) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 4 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neutrophil count increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procalcitonin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Red blood cell sedimentation rate increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reticulocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sars-cov-2 test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin b12 decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin d decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 2 (2) | 6 (8) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carbohydrate intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Folate deficiency (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 2 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 4 (10) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (4) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insulin resistance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin b complex deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin b12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (14) | 9 (11) | 1 (1) | 0 (0) | 3 (5) | 4 (4) | 1 (1) | 1 (1) | 3 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Axial spondyloarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (5) | 1 (1) | 0 (0) | 3 (3) | 4 (4) | 1 (1) | 2 (2) | 3 (3)
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chondropathy (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enthesopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femoroacetabular impingement (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (6) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/124 (1) | 0/88 (0) | 0/17 (0) | 0/11 (0) | 0/70 (0) | 0/54 (0) | 0/7 (0) | 0/21 (0) | 0/49 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Basal ganglia infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burning feet syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 10 (13) | 8 (8) | 0 (0) | 0 (0) | 3 (4) | 4 (4) | 0 (0) | 2 (4) | 11 (22)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (7)
Nerve compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ophthalmic migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Generalised anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersexuality (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Obsessive-compulsive disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stress (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Albuminuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract inflammation (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/163 (1) | 0/134 (0) | 0/12 (0) | 0/23 (0) | 0/68 (0) | 0/55 (0) | 0/11 (0) | 0/32 (0) | 0/57 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 1/124 (1) | 0/88 (0) | 0/17 (0) | 0/11 (0) | 0/70 (0) | 1/54 (1) | 0/7 (0) | 0/21 (0) | 1/49 (1)
Endometriosis (Reproductive system and breast disorders) | 0/124 (0) | 0/88 (0) | 0/17 (0) | 1/11 (2) | 0/70 (0) | 0/54 (0) | 0/7 (0) | 0/21 (0) | 0/49 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0/124 (0) | 0/88 (0) | 0/17 (0) | 0/11 (0) | 1/70 (1) | 0/54 (0) | 0/7 (0) | 0/21 (0) | 0/49 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0/124 (0) | 1/88 (1) | 0/17 (0) | 0/11 (0) | 0/70 (0) | 0/54 (0) | 0/7 (0) | 0/21 (0) | 0/49 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0/124 (0) | 0/88 (0) | 0/17 (0) | 0/11 (0) | 0/70 (0) | 1/54 (1) | 0/7 (0) | 0/21 (0) | 0/49 (0)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0/124 (0) | 0/88 (0) | 0/17 (0) | 0/11 (0) | 0/70 (0) | 0/54 (0) | 0/7 (0) | 1/21 (1) | 0/49 (0)
Pelvic fluid collection (Reproductive system and breast disorders) | 1/124 (1) | 0/88 (0) | 0/17 (0) | 0/11 (0) | 0/70 (0) | 0/54 (0) | 0/7 (0) | 0/21 (0) | 0/49 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 0/163 (0) | 0/134 (0) | 1/12 (1) | 0/23 (0) | 0/68 (0) | 0/55 (0) | 0/11 (0) | 0/32 (0) | 0/57 (0)
Prostatitis (Reproductive system and breast disorders) | 1/163 (1) | 0/134 (0) | 1/12 (1) | 0/23 (0) | 0/68 (0) | 0/55 (0) | 0/11 (0) | 0/32 (0) | 0/57 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/124 (0) | 0/88 (0) | 0/17 (0) | 0/11 (0) | 0/70 (0) | 0/54 (0) | 0/7 (0) | 1/21 (1) | 0/49 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0/124 (0) | 0/88 (0) | 0/17 (0) | 0/11 (0) | 0/70 (0) | 0/54 (0) | 0/7 (0) | 1/21 (1) | 0/49 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Choking sensation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Paranasal sinus inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Capillaritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukonychia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nodular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 8 (9) | 4 (5) | 0 (0) | 0 (0) | 5 (6) | 4 (5) | 1 (1) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sensitive skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urticaria papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Food contamination (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess drainage (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal fistula repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blepharoplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drainage (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dupuytren's contracture operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fistula repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoid operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileocolectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal anastomosis (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Intra-uterine contraceptive device insertion (Surgical and medical procedures) | 0/124 (0) | 0/88 (0) | 0/17 (0) | 0/11 (0) | 0/70 (0) | 0/54 (0) | 0/7 (0) | 0/21 (0) | 1/49 (1)
Keratomileusis (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laser therapy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liposuction (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mass excision (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device implantation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mole excision (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polypectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tenolysis (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Wisdom teeth removal (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brachiocephalic arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperaemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 4 (4)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Macroangiopathy (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2024-09-10): https://cdn.clinicaltrials.gov/large-docs/53/NCT04232553/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-10): https://cdn.clinicaltrials.gov/large-docs/53/NCT04232553/SAP_001.pdf